CLINICAL TRIAL: NCT03318718
Title: Paraspinal Muscle Relaxation in Spine Surgery: Comparison of the Effect of Neuromuscular Blocking Agent Rocuronium Between Extremity- and Paraspinal Musculature
Brief Title: Paraspinal Muscle Relaxation in Spine Surgery
Acronym: TOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOF
Record Dates: First submitted 2017-06-29; First posted 2017-10-24 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Paraspinal Muscle Relaxation in Spine Surgery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOF measurement (Experimental): TOF and MEP measurement after Anesthesia with non-depolarizing NMBA Rocuronium
  Interventions: Drug: Anesthesia with non-depolarizing NMBA Rocuronium; Diagnostic Test: TOF measurement; Diagnostic Test: MEP measurement

INTERVENTIONS:
Drug: Anesthesia with non-depolarizing NMBA Rocuronium — Non- depolarizing NMBA Rocuronium will be used until full paraspinal muscle Relaxation. Muscle relaxation during surgery will be performed using intraoperative boli intermediate duration non-depolarizing NMBA, rocuronium (0.3 mg/kg) until good surgical conditions are achieved.
Diagnostic Test: TOF measurement — TOF (Train-of-four) measurements will be performed at baseline 5 minutes after induction after the effect of succinylcholine will have run off. Moreover, TOF measurements will be performed 5 minutes after each rocuronium bolus
Diagnostic Test: MEP measurement — MEPs (motor evoked potentials) are routinely obtained after intubation and before surgery, then every 10min during the critical preparation and closing phases of surgery and every 5min during the correction phase. In addition MEPs will be measured after the administration of the NMBA rocuronium. Baseline values for amplitudes and latencies are obtained directly prior to the start of the correction phase of the surgery.

SUMMARY:
During anesthesia, neuromuscular blocking agents (NMBA) are routinely used for relaxation of muscles necessary for the conduction of the surgical procedure. Train-of-four (TOF) test is based on supramaximal stimulation of peripheral nerve resulting in four twitches: T1 to T4. The assessment of the NMBA blockade is performed routinely by measurement of the amplitude of compound muscle action potential (CMAP) and calculation of percentage of CMAP decrement from T1 to T4.

Train-of-four monitoring is routinely performed during spine surgery by stimulation of the ulnar nerve. Furthermore motor evoked potentials (MEPs) are routinely used in intraoperative neuromonitoring to assess the whole motor pathway from the cortical level down to the distal muscle. During anesthesia MEPs are routinely evoked by transcranial electrical stimulation with single or short train stimuli. In clinical practice even though full muscle relaxation of the hand by NMBA can be observed, utilizing the TOF test, remaining muscle tonus can be observed at the paraspinal musculature during spine surgery.

The goals of this study are to determine (1) if any differences between muscle relaxation of the hand and foot (measured by TOF test and MEPs) and MEPs of the paraspinal musculature occur; (2) how much more NMBA must be administered to achieve full muscle relaxation of the paraspinal musculature in comparison to the hand or foot.

DETAILED DESCRIPTION:
Muscle relaxation during surgery will be performed using intraoperative boli intermediate duration non-depolarizing NMBA, rocuronium (0.3 mg/kg) until TOF 0 at the hand is achieved. TOF measurements will be performed at baseline 5 minutes after induction. Moreover, TOF measurements will be performed 5 minutes after each rocuronium bolus. When TOF 0 at the hand is achieved the MEPs of the paraspinal musculature will be measured. When there is remaining muscle tonus of the paraspinal musculature another bolus of rocuronium is administered until no MEPs can be measured for the paraspinal musculature.

ELIGIBILITY:
Inclusion Criteria:

* All patients that will undergo spinal surgery with intraoperative neurophysiological Monitoring
* Age: 14 - 99 years

Exclusion Criteria:

* No intraoperative neurophysiological Monitoring
* Age <14 year
* prior neurological diseases or deficits that may affect safety of surgery/Intraoperative neuromonitoring
* No informed consent

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
assessment of NMBA blockade | during surgery
  assessment of the NMBA (neuromuscular blocking agent) blockade by measurement of the amplitude of compound muscle action potential (CMAP)
MEP | during surgery
  Motor evoked potentials (MEPs) are measured in hand, foot and paraspinal musculature
TOF | during surgery
  peak-to-peak amplitude of CMAP for each of 4 muscle contractions is measured. (supramaximal stimulation of peripheral nerve results in four twitches: T1 to T4)

SECONDARY OUTCOMES:
necessary administered amount of NMBA | during surgery
  Difference in the necessary administered amount of NMBA to achieve full muscle relaxation for hand and foot versus paraspinal musculature

CONTACTS AND LOCATIONS:
Overall Officials: Michael Betz, Dr.med., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Betz M, Aguirre J, Schubert M, Gotschi T, Huber B, Schupbach R, Brada M, Spirig JM, Farshad M. Hand or foot train-of-four tests and surgical site muscle relaxation assessed with multiple motor evoked potentials: A prospective observational study. Eur J Anaesthesiol. 2021 Aug 1;38(8):872-879. doi: 10.1097/EJA.0000000000001398. PMID 33259448